CLINICAL TRIAL: NCT06264362
Title: Developing a Nonpharmacological Pain Intervention for Community-dwelling Older Adults With Dementia
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Drexel University (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: K23AG081547 (NIH); 1K23AG081547-01 (NIH)
Record Dates: First submitted 2023-12-14; First posted 2024-02-20 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Pain, Chronic; Dementia, Mild; Mobility Limitation; Physical Disability; Osteo Arthritis Knee; Mild Cognitive Impairment
Keywords: pain; dementia; cognitive impairment; osteoarthritis; knee pain; memory
MeSH Terms: conditions — Chronic Pain; Dementia; Lymphoma, Follicular; Mobility Limitation; Cognitive Dysfunction; Pain; Osteoarthritis

STUDY DESIGN:
Intervention Model Description: In Phase 1 (not a clinical trial), 15 dyads and 15 clinicians will be interviewed (a dyad equals one person living with mild to very mild dementia and their care partner) to inform design of the intervention. In Phase 2 (a clinical trial), 20 people living with mild to very mild dementia will be treated with the new intervention. Their care partners may be involved in treatment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tailored Physical Activity Program for Pain (Experimental): Specific characteristics of the intervention delivered in Phase 2 will be based on the information gathered from stakeholders in Phase 1.
  Interventions: Behavioral: Tailored Physical Activity Program

INTERVENTIONS:
Behavioral: Tailored Physical Activity Program — Adaptation of physical activity as an intervention for pain management using the 3-Step Tailored Approach: assessing in Step 1 the Person Living with Dementia (PLWD), in Step 2 the Environment, and in Step 3 the Caregiver. With this approach, traditional exercises can be adapted to 1) functional activities (e.g., stair climbing) that are tailored to the interests (e.g., dancing, boxing) and preserved abilities of PLWD; 2) preferred and well-tolerated environments (e.g., home); and 3) account for extent and type of interventionist and caregiver involvement.

SUMMARY:
The purpose of this study is to develop an exercise treatment program for knee osteoarthritis that works well for people with memory problems. This study will include two parts. Participants can choose to participate in either or both parts.

In Part 1 (not a clinical trial) - The investigators are inviting the following people to participate in an interview:

1. Individuals aged 60 years or older who do not live in a nursing home and have both memory issues and knee pain.
2. Care partners of people with knee pain and memory issues. A care partner can be a family member or friend who helps regularly.
3. Clinicians (exercise physiologists or rehabilitation therapists like physical and occupational therapists) who have worked with older adults with memory issues and knee pain.

The goal of these interviews is to learn from the experiences of people with memory issues and knee pain and those who care for them. From these interviews, the investigators hope to design a non-drug, tailored physical activity program that will be interesting and helpful in managing knee pain for older adults with memory problems.

For people with memory problems and knee pain and their care partners: The investigators will ask some questions to determine eligibility to participate in the study.

Those who qualify for the study will be invited to participate in an interview that could be completed online or in person (Philadelphia, PA). The interview could last up to 90 minutes (1 and a half hours) and can be completed as one or multiple sessions.

For clinicians: Participants will engage in a 90-minute focus group with other clinicians where lunch will be served if in person. Those participating in an online focus group will receive a gift card equal to the value of lunch.

In Part 2 (a clinical trial) - The program developed in Part 1 will be tested. The program will be physical activity-based. Specific program details for part 2 will be provided as they emerge. Participants can choose to sign up for either or both parts. Signing up for Part 1 does not mean participants have to sign up for Part 2.

Please contact us for any questions.

DETAILED DESCRIPTION:
Chronic musculoskeletal pain, specifically osteoarthritis (OA) of the knee, is common among community-dwelling people living with memory issues and associated with cascading negative consequences on physical function limitations, quality of life decline, and caregiver burden; however, few beneficial and appropriate treatment options exist. This study seeks to use evidence, theory, and stakeholder input to design an exercise-based intervention for knee OA pain management tailored to the interests, preserved abilities, and biopsychosocial-environmental needs of community-dwelling older adults with mild to very mild dementia. Findings from K23 research will yield a nonpharmacological intervention prototype and delivery parameters that will inform a future efficacy study and have a strong potential for preserving or improving the quality of life of community-dwelling older adults with dementia and OA.

ELIGIBILITY:
Inclusion Criteria for people living with dementia:

* Age 60 or older
* Speaks English
* Mild/Very Mild dementia
* Knee pain lasting ≥ 3 months, potentially related to arthritis
* Knee pain is at least 2 out of 10 on average.

Exclusion Criteria for people living with dementia:

* Reside in long term care facility
* Unable or unwilling to consent
* Has a condition with a life expectancy of less than 1-year
* No care partner who is also willing to participate
* Recent changes to pain or psychotropic medications in the last 60 days
* Recent knee surgery in the last 1-year
* Has a condition that contraindicates exercise (Phase 2 only)
* Currently receiving rehab services (Phase 2 only)

For care partners:

* No sex, gender, or age criteria
* Has known person living with dementia ≥ 1 year
* Speaks English
* Able and willing to consent, including being recorded

For clinicians:

* No sex, gender, or age criteria
* Speaks English
* Has ≥ 2 years of experience working with community-dwelling people with dementia and pain
* Able and willing to consent, including being recorded

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-06-02 (Estimated); Primary Completion 2027-03-31 (Estimated); Study Completion 2027-05-01 (Estimated)

PRIMARY OUTCOMES:
Program parameters | Day 1
  Qualitative interviews to determine preferred program parameters.
Program parameters | Day 1
  Focus groups of clinicians to determine preferred program parameters.
Feasibility of Intervention Measure | At study completion, an average of 8 weeks
  The Feasibility of Intervention Measure is a standardized 4-question self-reported outcome measure to assess feasibility. Each item is scored on a 5-point scale, where 1 = completely disagree, 2 = disagree, 3 = neither agree or disagree, 4 = agree, 5 = completely agree. The responses are summed and range between 5 to 20, with higher scores indicating greater feasibility. A score of 16 or greater suggests the program is feasible, 15 to 9 indicates the program may be feasible, and a score of 8 or less suggests the program is not feasible.
Perception of program | At study completion, an average of 8 weeks
  Qualitative Interview of all who participated in the program to determine components of the intervention prototype that needs revising

SECONDARY OUTCOMES:
Numeric Pain Score | Through study completion, an average of 8 weeks.
  A self-reported pain measurement ranging from 0 (no pain) to 10 (worst pain). A high score indicates more pain.
Zarit Burden Interview-Short Form | At study completion, an average of 8 weeks
  Zarit Burden Interview-Short Form is a12-item questionnaire to assess the burden of caregiving using a 5-point scale where 0 (never) to 4 (almost always). Scores are summed, ranging from 0-48, where a higher score indicates a greater caregiver burden.

CONTACTS AND LOCATIONS:
Overall Officials: Annalisa Na, PT, PhD, Principal Investigator — Drexel University
Locations (1):
- Drexel University, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Innes KE, Sambamoorthi U. The Association of Osteoarthritis and Related Pain Burden to Incident Alzheimer's Disease and Related Dementias: A Retrospective Cohort Study of U.S. Medicare Beneficiaries. J Alzheimers Dis. 2020;75(3):789-805. doi: 10.3233/JAD-191311. PMID 32333589
- [Background] Hunt LJ, Covinsky KE, Yaffe K, Stephens CE, Miao Y, Boscardin WJ, Smith AK. Pain in Community-Dwelling Older Adults with Dementia: Results from the National Health and Aging Trends Study. J Am Geriatr Soc. 2015 Aug;63(8):1503-11. doi: 10.1111/jgs.13536. Epub 2015 Jul 22. PMID 26200445
- [Background] Sverdrup K, Bergh S, Selbaek G, Benth JS, Roen IM, Husebo B, Tangen GG. Trajectories of physical performance in nursing home residents with dementia. Aging Clin Exp Res. 2020 Dec;32(12):2603-2610. doi: 10.1007/s40520-020-01499-y. Epub 2020 Feb 14. PMID 32060802
- [Background] Tanaka H, Nagata Y, Ishimaru D, Ogawa Y, Fukuhara K, Nishikawa T. Clinical factors associated with activities of daily living and their decline in patients with severe dementia. Psychogeriatrics. 2020 May;20(3):327-336. doi: 10.1111/psyg.12502. Epub 2019 Dec 28. PMID 31883310
- [Background] APTA Geriatrics Combined Sections Meeting 2022 Poster Abstracts. J Geriatr Phys Ther. 2022 Jan-Mar 01;45(1):E16-E77. doi: 10.1519/JPT.0000000000000336. No abstract available. PMID 34928240
- [Background] Gitlin LN, Arthur P, Piersol C, Hessels V, Wu SS, Dai Y, Mann WC. Targeting Behavioral Symptoms and Functional Decline in Dementia: A Randomized Clinical Trial. J Am Geriatr Soc. 2018 Feb;66(2):339-345. doi: 10.1111/jgs.15194. Epub 2017 Nov 28. PMID 29192967
- [Background] Whitlock EL, Diaz-Ramirez LG, Glymour MM, Boscardin WJ, Covinsky KE, Smith AK. Association Between Persistent Pain and Memory Decline and Dementia in a Longitudinal Cohort of Elders. JAMA Intern Med. 2017 Aug 1;177(8):1146-1153. doi: 10.1001/jamainternmed.2017.1622. PMID 28586818
- [Background] Hodgson N, Gitlin LN, Huang J. The influence of sleep disruption and pain perception on indicators of quality of life in individuals living with dementia at home. Geriatr Nurs. 2014 Sep-Oct;35(5):394-8. doi: 10.1016/j.gerinurse.2014.08.005. Epub 2014 Sep 2. PMID 25193739
- [Background] Monroe TB, Misra SK, Habermann RC, Dietrich MS, Cowan RL, Simmons SF. Pain reports and pain medication treatment in nursing home residents with and without dementia. Geriatr Gerontol Int. 2014 Jul;14(3):541-8. doi: 10.1111/ggi.12130. Epub 2013 Sep 11. PMID 24020433
- [Background] Rundell SD, Phelan EA, Patel KV, Jones BL, Marcum ZA. Longitudinal Patterns of Pain Reporting Among Community-dwelling Older Adults. Clin J Pain. 2020 Dec;36(12):912-922. doi: 10.1097/AJP.0000000000000874. PMID 32841970
- [Background] 2020 Alzheimer's disease facts and figures. Alzheimers Dement. 2020 Mar 10. doi: 10.1002/alz.12068. Online ahead of print. PMID 32157811
- [Background] AGS clinical practice guidelines: the management of chronic pain in older persons. Geriatrics. 1998 Oct;53 Suppl 3:S6-7. No abstract available. PMID 9826951
- [Background] Bullock L, Bedson J, Jordan JL, Bartlam B, Chew-Graham CA, Campbell P. Pain assessment and pain treatment for community-dwelling people with dementia: A systematic review and narrative synthesis. Int J Geriatr Psychiatry. 2019 Jun;34(6):807-821. doi: 10.1002/gps.5078. Epub 2019 Apr 8. PMID 30724409
- [Background] Bullock L, Chew-Graham CA, Bedson J, Bartlam B, Campbell P. The challenge of pain identification, assessment, and management in people with dementia: a qualitative study. BJGP Open. 2020 Jun 23;4(2):bjgpopen20X101040. doi: 10.3399/bjgpopen20X101040. Print 2020. PMID 32457099
- [Background] Corbett A, Nunez KM, Smeaton E, Testad I, Thomas AJ, Closs SJ, Briggs M, Clifton L, Gjestsen MT, Lawrence V. The landscape of pain management in people with dementia living in care homes: a mixed methods study. Int J Geriatr Psychiatry. 2016 Dec;31(12):1354-1370. doi: 10.1002/gps.4445. Epub 2016 Feb 21. PMID 26898542
- [Background] Gagliese L, Gauthier LR, Narain N, Freedman T. Pain, aging and dementia: Towards a biopsychosocial model. Prog Neuropsychopharmacol Biol Psychiatry. 2018 Dec 20;87(Pt B):207-215. doi: 10.1016/j.pnpbp.2017.09.022. Epub 2017 Sep 22. PMID 28947182
- [Background] American Geriatrics Society Panel on Exercise and Osteoarthritis. Exercise prescription for older adults with osteoarthritis pain: consensus practice recommendations. A supplement to the AGS Clinical Practice Guidelines on the management of chronic pain in older adults. J Am Geriatr Soc. 2001 Jun;49(6):808-23. doi: 10.1046/j.1532-5415.2001.00496.x. No abstract available. PMID 11480416
- [Background] Brown GA. AAOS clinical practice guideline: treatment of osteoarthritis of the knee: evidence-based guideline, 2nd edition. J Am Acad Orthop Surg. 2013 Sep;21(9):577-9. doi: 10.5435/JAAOS-21-09-577. No abstract available. PMID 23996989
- [Background] Kolasinski SL, Neogi T, Hochberg MC, Oatis C, Guyatt G, Block J, Callahan L, Copenhaver C, Dodge C, Felson D, Gellar K, Harvey WF, Hawker G, Herzig E, Kwoh CK, Nelson AE, Samuels J, Scanzello C, White D, Wise B, Altman RD, DiRenzo D, Fontanarosa J, Giradi G, Ishimori M, Misra D, Shah AA, Shmagel AK, Thoma LM, Turgunbaev M, Turner AS, Reston J. 2019 American College of Rheumatology/Arthritis Foundation Guideline for the Management of Osteoarthritis of the Hand, Hip, and Knee. Arthritis Rheumatol. 2020 Feb;72(2):220-233. doi: 10.1002/art.41142. Epub 2020 Jan 6. PMID 31908163
- [Background] Gitlin LN, Hodgson NA. Better Living with Dementia: Implications for Individuals, Families, Communities, and Societies. Elsevier Academic Press; 2018.
- [Background] Morone NE, Abebe KZ, Morrow LA, Weiner DK. Pain and decreased cognitive function negatively impact physical functioning in older adults with knee osteoarthritis. Pain Med. 2014 Sep;15(9):1481-7. doi: 10.1111/pme.12483. Epub 2014 Jul 8. PMID 25040845
- [Background] Coronado RA, Albers HE, Allen JL, Clarke RG, Estrada VA, Simon CB, Galloway RV, Fisher SR. Pain-Reducing Effects of Physical Therapist-Delivered Interventions: A Systematic Review of Randomized Trials Among Older Adults With Dementia. J Geriatr Phys Ther. 2020 Jul/Sep;43(3):159-169. doi: 10.1519/JPT.0000000000000235. PMID 30998563
- [Background] Pieper MJ, van Dalen-Kok AH, Francke AL, van der Steen JT, Scherder EJ, Husebo BS, Achterberg WP. Interventions targeting pain or behaviour in dementia: a systematic review. Ageing Res Rev. 2013 Sep;12(4):1042-55. doi: 10.1016/j.arr.2013.05.002. Epub 2013 May 28. PMID 23727161
- [Background] Pu L, Moyle W, Jones C, Todorovic M. Psychosocial interventions for pain management in older adults with dementia: A systematic review of randomized controlled trials. J Adv Nurs. 2019 Aug;75(8):1608-1620. doi: 10.1111/jan.13929. Epub 2019 Jan 15. PMID 30537124
- [Background] Gibson SJ. IASP global year against pain in older persons: highlighting the current status and future perspectives in geriatric pain. Expert Rev Neurother. 2007 Jun;7(6):627-35. doi: 10.1586/14737175.7.6.627. PMID 17563246
- [Background] Bradt J, Burns DS, Creswell JW. Mixed methods research in music therapy research. J Music Ther. 2013 Summer;50(2):123-48. doi: 10.1093/jmt/50.2.123. PMID 24156190
- [Background] The management of chronic pain in older persons: AGS Panel on Chronic Pain in Older Persons. American Geriatrics Society. J Am Geriatr Soc. 1998 May;46(5):635-51. doi: 10.1111/j.1532-5415.1998.tb01084.x. No abstract available. PMID 9588381
- [Background] Achterberg W, Lautenbacher S, Husebo B, Erdal A, Herr K. Pain in dementia. Pain Rep. 2019 Dec 25;5(1):e803. doi: 10.1097/PR9.0000000000000803. eCollection 2020 Jan-Feb. PMID 32072098
- [Background] Cohen-Mansfield J. The relationship between different pain assessments in dementia. Alzheimer Dis Assoc Disord. 2008 Jan-Mar;22(1):86-93. doi: 10.1097/WAD.0b013e3181630b5c. PMID 18317252
- [Background] Hodgson N, Gitlin LN, Winter L, Hauck WW. Caregiver's perceptions of the relationship of pain to behavioral and psychiatric symptoms in older community-residing adults with dementia. Clin J Pain. 2014 May;30(5):421-7. doi: 10.1097/AJP.0000000000000018. PMID 24281271
- [Background] de Souto Barreto P, Denormandie P, Lepage B, Armaingaud D, Rapp T, Chauvin P, Vellas B, Rolland Y. Effects of a long-term exercise programme on functional ability in people with dementia living in nursing homes: Research protocol of the LEDEN study, a cluster randomised controlled trial. Contemp Clin Trials. 2016 Mar;47:289-95. doi: 10.1016/j.cct.2016.02.004. Epub 2016 Feb 13. PMID 26883281
- [Background] Canavan PK, Cahalin LP, Lowe S, Fitzpatrick D, Harris M, Plummer-D'Amato P. Managing gait disorders in older persons residing in nursing homes: a review of literature. J Am Med Dir Assoc. 2009 May;10(4):230-7. doi: 10.1016/j.jamda.2009.02.008. PMID 19426938
- [Background] de Souto Barreto P, Cesari M, Denormandie P, Armaingaud D, Vellas B, Rolland Y. Exercise or Social Intervention for Nursing Home Residents with Dementia: A Pilot Randomized, Controlled Trial. J Am Geriatr Soc. 2017 Sep;65(9):E123-E129. doi: 10.1111/jgs.14947. Epub 2017 May 19. PMID 28542742
- [Background] Goncalves AC, Demain S, Samuel D, Marques A. Physical activity for people living with dementia: carer outcomes and side effects from the perspectives of professionals and family carers. Aging Clin Exp Res. 2021 May;33(5):1267-1274. doi: 10.1007/s40520-020-01636-7. Epub 2020 Jul 3. PMID 32621269
- [Background] Hauer K, Lemke NC, Werner C, Wiloth S. Transferability and Sustainability of Effects of Dual-Task Training in Patients with Dementia. Journal: Conference Abstract. Eur Geriatr Med. 2018;9:S248-S249.
- [Background] Lam FMH, Liao LR, Kwok TCY, Pang MYC. Effects of adding whole-body vibration to routine day activity program on physical functioning in elderly with mild or moderate dementia: a randomized controlled trial. Int J Geriatr Psychiatry. 2018 Jan;33(1):21-30. doi: 10.1002/gps.4662. Epub 2017 Jan 17. PMID 28094873
- [Background] Larmer PJ, Reay ND, Aubert ER, Kersten P. Systematic review of guidelines for the physical management of osteoarthritis. Arch Phys Med Rehabil. 2014 Feb;95(2):375-89. doi: 10.1016/j.apmr.2013.10.011. Epub 2013 Nov 1. PMID 24184307
- [Background] Durmus D, Alayli G, Canturk F. Effects of quadriceps electrical stimulation program on clinical parameters in the patients with knee osteoarthritis. Clin Rheumatol. 2007 May;26(5):674-8. doi: 10.1007/s10067-006-0358-3. Epub 2006 Aug 1. PMID 16897119
- [Background] Weiner BJ, Lewis CC, Stanick C, Powell BJ, Dorsey CN, Clary AS, Boynton MH, Halko H. Psychometric assessment of three newly developed implementation outcome measures. Implement Sci. 2017 Aug 29;12(1):108. doi: 10.1186/s13012-017-0635-3. PMID 28851459
- [Background] Achterberg WP, Pieper MJ, van Dalen-Kok AH, de Waal MW, Husebo BS, Lautenbacher S, Kunz M, Scherder EJ, Corbett A. Pain management in patients with dementia. Clin Interv Aging. 2013;8:1471-82. doi: 10.2147/CIA.S36739. Epub 2013 Nov 1. PMID 24204133
- [Background] Gitlin LN, Hodgson N, Piersol CV, Hess E, Hauck WW. Correlates of quality of life for individuals with dementia living at home: the role of home environment, caregiver, and patient-related characteristics. Am J Geriatr Psychiatry. 2014 Jun;22(6):587-97. doi: 10.1016/j.jagp.2012.11.005. Epub 2013 Jul 25. PMID 23890928
- [Background] Bartholomew LK, Parcel GS, Kok G. Intervention mapping: a process for developing theory- and evidence-based health education programs. Health Educ Behav. 1998 Oct;25(5):545-63. doi: 10.1177/109019819802500502. PMID 9768376
- [Background] Booth V, Hood-Moore V, Hancox JE, Logan P, Robinson KR. Systematic scoping review of frameworks used to develop rehabilitation interventions for older adults. BMJ Open. 2019 Feb 22;9(2):e024185. doi: 10.1136/bmjopen-2018-024185. PMID 30798309
- [Background] Craig P, Dieppe P, Macintyre S, Michie S, Nazareth I, Petticrew M. Developing and evaluating complex interventions: the new Medical Research Council guidance. Int J Nurs Stud. 2013 May;50(5):587-92. doi: 10.1016/j.ijnurstu.2012.09.010. Epub 2012 Nov 15. No abstract available. PMID 23159157
- [Background] O'Cathain A, Croot L, Duncan E, Rousseau N, Sworn K, Turner KM, Yardley L, Hoddinott P. Guidance on how to develop complex interventions to improve health and healthcare. BMJ Open. 2019 Aug 15;9(8):e029954. doi: 10.1136/bmjopen-2019-029954. PMID 31420394
- [Background] Skivington K, Matthews L, Simpson SA, Craig P, Baird J, Blazeby JM, Boyd KA, Craig N, French DP, McIntosh E, Petticrew M, Rycroft-Malone J, White M, Moore L. A new framework for developing and evaluating complex interventions: update of Medical Research Council guidance. BMJ. 2021 Sep 30;374:n2061. doi: 10.1136/bmj.n2061. PMID 34593508
- [Background] Creswell JWPCVL. Designing and Conducting Mixed Methods Research. 2018.
- [Background] Billingham SA, Whitehead AL, Julious SA. An audit of sample sizes for pilot and feasibility trials being undertaken in the United Kingdom registered in the United Kingdom Clinical Research Network database. BMC Med Res Methodol. 2013 Aug 20;13:104. doi: 10.1186/1471-2288-13-104. PMID 23961782
- [Background] Gitlin LN, Marx KA, Alonzi D, Kvedar T, Moody J, Trahan M, Van Haitsma K. Feasibility of the Tailored Activity Program for Hospitalized (TAP-H) Patients With Behavioral Symptoms. Gerontologist. 2017 Jun;57(3):575-584. doi: 10.1093/geront/gnw052. Epub 2016 Apr 13. PMID 27076056
- [Background] Browne RH. On the use of a pilot sample for sample size determination. Stat Med. 1995 Sep 15;14(17):1933-40. doi: 10.1002/sim.4780141709. PMID 8532986
- [Background] Eldridge SM, Chan CL, Campbell MJ, Bond CM, Hopewell S, Thabane L, Lancaster GA; PAFS consensus group. CONSORT 2010 statement: extension to randomised pilot and feasibility trials. BMJ. 2016 Oct 24;355:i5239. doi: 10.1136/bmj.i5239. PMID 27777223
- [Background] Eldridge SM, Lancaster GA, Campbell MJ, Thabane L, Hopewell S, Coleman CL, Bond CM. Defining Feasibility and Pilot Studies in Preparation for Randomised Controlled Trials: Development of a Conceptual Framework. PLoS One. 2016 Mar 15;11(3):e0150205. doi: 10.1371/journal.pone.0150205. eCollection 2016. PMID 26978655
- [Background] Thabane L, Hopewell S, Lancaster GA, Bond CM, Coleman CL, Campbell MJ, Eldridge SM. Methods and processes for development of a CONSORT extension for reporting pilot randomized controlled trials. Pilot Feasibility Stud. 2016 May 20;2:25. doi: 10.1186/s40814-016-0065-z. eCollection 2016. PMID 27965844
- [Background] Kim YS, Park JM, Moon YS, Han SH. Assessment of pain in the elderly: A literature review. Natl Med J India. 2017 Jul-Aug;30(4):203-207. doi: 10.4103/0970-258X.218673. PMID 29162753
- [Background] Herr K. Pain assessment in cognitively impaired older adults. Am J Nurs. 2002 Dec;102(12):65-7. doi: 10.1097/00000446-200212000-00020. No abstract available. PMID 12473932
- [Background] Herr KA, Mobily PR, Kohout FJ, Wagenaar D. Evaluation of the Faces Pain Scale for use with the elderly. Clin J Pain. 1998 Mar;14(1):29-38. doi: 10.1097/00002508-199803000-00005. PMID 9535311
- [Background] Van Rickstal R, Vleminck A, Engelborghs S, Versijpt J, Van den Block L. A qualitative study with people with young-onset dementia and their family caregivers on advance care planning: A holistic, flexible, and relational approach is recommended. Palliat Med. 2022 Jun;36(6):964-975. doi: 10.1177/02692163221090385. Epub 2022 Apr 26. PMID 35470742
- [Background] Hartmann J, Rossmeier C, Riedl L, Dorn B, Fischer J, Slawik T, Fleischhaker M, Hartmann F, Egert-Schwender S, Kehl V, Haller B, Schneider-Schelte H, Dinkel A, Jox RJ, Diehl-Schmid J. Quality of Life in Advanced Dementia with Late Onset, Young Onset, and Very Young Onset. J Alzheimers Dis. 2021;80(1):283-297. doi: 10.3233/JAD-201302. PMID 33523011
- [Background] Kuruppu DK, Matthews BR. Young-onset dementia. Semin Neurol. 2013 Sep;33(4):365-85. doi: 10.1055/s-0033-1359320. Epub 2013 Nov 14. PMID 24234358
- [Background] Frank L, Shubeck E, Schicker M, Webb T, Maslow K, Gitlin L, Hummel CH, Kaplan EK, LeBlanc B, Marquez M, Nicholson B, O'Brien G, Phillips L, Van Buren B, Epstein-Lubow G. Contributions of Persons Living With Dementia to Scientific Research Meetings. Results From the National Research Summit on Care, Services, and Supports for Persons With Dementia and Their Caregivers. Am J Geriatr Psychiatry. 2020 Apr;28(4):421-430. doi: 10.1016/j.jagp.2019.10.014. Epub 2019 Oct 28. PMID 31784409
- [Background] Frank L, Shubeck E, Schicker M, Webb T, Maslow K, Gitlin L, Hummel CH, Kaplan EK, LeBlanc B, Marquez M, Nicholson BP, O'Brien G, Phillips L, Van Buren B, Epstein-Lubow G. The Experiences of Persons Living with Dementia Planning for a Dementia Research Meeting. Lessons Learned From the National Research Summit on Care, Services, and Supports for Persons With Dementia and Their Caregivers. Am J Geriatr Psychiatry. 2020 Apr;28(4):434-442. doi: 10.1016/j.jagp.2019.10.015. Epub 2019 Oct 28. PMID 31767451
- [Background] Elo S, Kyngas H. The qualitative content analysis process. J Adv Nurs. 2008 Apr;62(1):107-15. doi: 10.1111/j.1365-2648.2007.04569.x. PMID 18352969
- [Background] Moser A, Korstjens I. Series: Practical guidance to qualitative research. Part 3: Sampling, data collection and analysis. Eur J Gen Pract. 2018 Dec;24(1):9-18. doi: 10.1080/13814788.2017.1375091. Epub 2017 Dec 4. PMID 29199486
- [Background] Braun V, Clarke V. Successful Qualitative Research: A Practical Guide for Beginners. SAGE Publications; 2013.
- [Background] Fugard AJB, Potts HWW. Supporting Thinking on Sample Sizes for Thematic Analyses: A Quantitative Tool. International Journal of Social Research Methodology. 2015/11/02 2015;18(6):669-684.
- [Background] Guest G, Namey E, Chen M. A simple method to assess and report thematic saturation in qualitative research. PLoS One. 2020 May 5;15(5):e0232076. doi: 10.1371/journal.pone.0232076. eCollection 2020. PMID 32369511
- [Background] Matthews KA, Xu W, Gaglioti AH, Holt JB, Croft JB, Mack D, McGuire LC. Racial and ethnic estimates of Alzheimer's disease and related dementias in the United States (2015-2060) in adults aged >/=65 years. Alzheimers Dement. 2019 Jan;15(1):17-24. doi: 10.1016/j.jalz.2018.06.3063. Epub 2018 Sep 19. PMID 30243772
- [Background] Korstjens I, Moser A. Series: Practical guidance to qualitative research. Part 4: Trustworthiness and publishing. Eur J Gen Pract. 2018 Dec;24(1):120-124. doi: 10.1080/13814788.2017.1375092. Epub 2017 Dec 5. PMID 29202616
- [Background] Gitlin LN, Kales HC, Lyketsos CG. Nonpharmacologic management of behavioral symptoms in dementia. JAMA. 2012 Nov 21;308(19):2020-9. doi: 10.1001/jama.2012.36918. PMID 23168825
- [Background] Gitlin LN, Winter L, Dennis MP, Hodgson N, Hauck WW. A biobehavioral home-based intervention and the well-being of patients with dementia and their caregivers: the COPE randomized trial. JAMA. 2010 Sep 1;304(9):983-91. doi: 10.1001/jama.2010.1253. PMID 20810376
- [Background] Nunan D, Aronson J, Bankhead C. Catalogue of bias: attrition bias. BMJ Evid Based Med. 2018 Feb;23(1):21-22. doi: 10.1136/ebmed-2017-110883. PMID 29367321
- [Background] Finch TL, Girling M, May CR, et al. Implementation Measure Based on Normalization Process Theory. [Measurement Instrument]. http://www.normalizationprocess.org.
- [Background] Finch TL, Girling M, May CR, Mair FS, Murray E, Treweek S, McColl E, Steen IN, Cook C, Vernazza CR, Mackintosh N, Sharma S, Barbery G, Steele J, Rapley T. Improving the normalization of complex interventions: part 2 - validation of the NoMAD instrument for assessing implementation work based on normalization process theory (NPT). BMC Med Res Methodol. 2018 Nov 15;18(1):135. doi: 10.1186/s12874-018-0591-x. PMID 30442094
- [Background] Rapley T, Girling M, Mair FS, Murray E, Treweek S, McColl E, Steen IN, May CR, Finch TL. Improving the normalization of complex interventions: part 1 - development of the NoMAD instrument for assessing implementation work based on normalization process theory (NPT). BMC Med Res Methodol. 2018 Nov 15;18(1):133. doi: 10.1186/s12874-018-0590-y. PMID 30442093
- [Background] Zwakhalen S, Docking RE, Gnass I, Sirsch E, Stewart C, Allcock N, Schofield P. Pain in older adults with dementia : A survey across Europe on current practices, use of assessment tools, guidelines and policies. Schmerz. 2018 Oct;32(5):364-373. doi: 10.1007/s00482-018-0290-x. PMID 29931391
- [Background] Liu JY, Briggs M, Closs SJ. The psychometric qualities of four observational pain tools (OPTs) for the assessment of pain in elderly people with osteoarthritic pain. J Pain Symptom Manage. 2010 Oct;40(4):582-98. doi: 10.1016/j.jpainsymman.2010.02.022. Epub 2010 Aug 8. PMID 20692806
- [Background] Warden V, Hurley AC, Volicer L. Development and psychometric evaluation of the Pain Assessment in Advanced Dementia (PAINAD) scale. J Am Med Dir Assoc. 2003 Jan-Feb;4(1):9-15. doi: 10.1097/01.JAM.0000043422.31640.F7. PMID 12807591
- [Background] Bentur N, Cohen-Mansfield J, Radomyslsky Z. Is Pain Assessment of Community-Dwelling Persons With Advanced Dementia by Family and Paid Care Workers Feasible? J Pain Symptom Manage. 2021 May;61(5):1028-1034. doi: 10.1016/j.jpainsymman.2020.11.004. Epub 2020 Nov 10. PMID 33186731
- [Background] Lewis CC, Weiner BJ, Stanick C, Fischer SM. Advancing implementation science through measure development and evaluation: a study protocol. Implement Sci. 2015 Jul 22;10:102. doi: 10.1186/s13012-015-0287-0. PMID 26197880
- [Background] Creswell JW, Klassen AC, Plano Clark VL, Smith KC. Best Practices for Mixed Methods Research in the Health Sciences. Bethesda (Maryland): National Institutes of Health. 2011;2013:541-545.
- [Background] Eldridge SM, Chan CL, Campbell MJ, Bond CM, Hopewell S, Thabane L, Lancaster GA; PAFS consensus group. CONSORT 2010 statement: extension to randomised pilot and feasibility trials. Pilot Feasibility Stud. 2016 Oct 21;2:64. doi: 10.1186/s40814-016-0105-8. eCollection 2016. PMID 27965879
- [Background] Schulz KF, Grimes DA. Sample size slippages in randomised trials: exclusions and the lost and wayward. Lancet. 2002 Mar 2;359(9308):781-5. doi: 10.1016/S0140-6736(02)07882-0. PMID 11888606
- [Background] Na A, Buchanan TS. Validating Wearable Sensors Using Self-Reported Instability among Patients with Knee Osteoarthritis. PM R. 2021 Feb;13(2):119-127. doi: 10.1002/pmrj.12393. Epub 2020 Aug 12. PMID 32358908
- [Background] Na A, Buchanan TS. Self-reported walking difficulty and knee osteoarthritis influences limb dynamics and muscle co-contraction during gait. Hum Mov Sci. 2019 Apr;64:409-419. doi: 10.1016/j.humov.2018.11.002. Epub 2018 Nov 15. PMID 30448202
- [Background] Na A, Piva SR, Buchanan TS. Influences of knee osteoarthritis and walking difficulty on knee kinematics and kinetics. Gait Posture. 2018 Mar;61:439-444. doi: 10.1016/j.gaitpost.2018.01.025. Epub 2018 Feb 2. PMID 29477961
- [Background] Na A, Jansky L, Gugala Z. Clinical Characteristics of Patients with Type 2 Diabetes Mellitus Receiving a Primary Total Knee or Hip Arthroplasty. J Diabetes Res. 2019 Nov 19;2019:9459206. doi: 10.1155/2019/9459206. eCollection 2019. PMID 31828171
- [Background] Na A, Oppermann LM, Jupiter DC, Lindsey RW, Coronado RA. Diabetes Mellitus Blunts the Symptoms, Physical Function, and Health-Related Quality of Life Benefits of Total Knee Arthroplasty: A Systematic Review With Meta-analysis of Data From More Than 17 000 Patients. J Orthop Sports Phys Ther. 2021 Jun;51(6):269-280. doi: 10.2519/jospt.2021.9515. Epub 2021 Apr 19. PMID 33870736
- [Background] Na A, Middleton A, Haas A, Graham JE, Ottenbacher KJ. Impact of Diabetes on 90-Day Episodes of Care After Elective Total Joint Arthroplasty Among Medicare Beneficiaries. J Bone Joint Surg Am. 2020 Dec 16;102(24):2157-2165. doi: 10.2106/JBJS.20.00203. PMID 33093299
- [Background] Na A, Richburg K, Gugala Z. Clinical Considerations for Return to Driving a Car following a Total Knee or Hip Arthroplasty: A Systematic Review. Biomed Res Int. 2020 Jul 6;2020:8921892. doi: 10.1155/2020/8921892. eCollection 2020. PMID 32724816